CLINICAL TRIAL: NCT00825448
Title: Impact for Care for Patients With Alcohol Addiction and Treated for ORL Cancer
Brief Title: Alcohol Addiction and Otorhinolaryngology Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department of Clinical Research and Innovation (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor-Investigator, Department of Clinical Research and Innovation, Department of Clinical Research and Innovation (drc), Centre Hospitalier Universitaire de Nice
Organization: Centre Hospitalier Universitaire de Nice (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008-A00634-51
Record Dates: First submitted 2009-01-20; First posted 2009-01-21 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2011-12

CONDITIONS: Cancer of the Upper Aero-digestive Tract; Alcoholism
Keywords: alcohol addiction
MeSH Terms: conditions — Alcoholism | interventions — Hospitalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): patient in hospital a week before the date of surgery for the treatment of his addiction alcohol
  Interventions: Procedure: Hospitalization for a week
- 1 (No Intervention): no treatment of his addiction alcohol during a week before the date of surgery

INTERVENTIONS:
Procedure: Hospitalization for a week — Patient in hospital a week before the date of surgery for the treatment of their addiction to alcohol (alcohol weaning)
  Arms: 2

SUMMARY:
The aim of the study is to compare the hospitalisation period in ORL surgery for two groups of patients. One of them will be treated for alcohol addiction to weaning them before the surgery ORL. The other group will be treated with usual methods.

DETAILED DESCRIPTION:
Alcohol, associated or not associated with tobacco, is known to increase the incidence of ORL cancer. So, in fact many patients perform their ORL surgery operation in spite of their alcohol addiction.

Many studies showed that a post surgery weaning syndrome increases morbidity and mortality.

So our study will focuses on the benefits of pre surgery medical weaning program.

The protocol is an open randomised, prospective study. The patient will be divided in two groups. In one hand, the first group is designed as "treated" will get alcohol weaning in the hospital alcohol department. The patient will be hospitalized during one week before the ORL surgery.

During this hospitalisation, the patient will receive medicinal treatment, medical follow-up and psychological counselling.

In the other hand, the second group designed as "control group" will be hospitalized directly in ORL surgery department. The patient will be received a treatment for alcohol weaning according to their symptom.

After their hospitalisation, the treated group will be followed-up regularly for their alcohol addiction either in support group or in individual counselling. The control group will be followed-up with the usual method in the ORL surgery department.

The expected result is to improve the care for patients with alcohol addiction and who must have an ORL surgery reducing the hospitalisation duration, the level of post operative complication and increasing the abstinence level. 115 patients will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years, male or female
* Clinically and histologically verified ORL cancer required surgery
* Patient with alcohol addiction
* Men must consume 21 glasses of wine a week
* Women must consume 14 glasses of wine a week
* CPAM affiliation
* Able to give written informed consent to participate in the study

Exclusion Criteria:

* Inability to give informed consent
* Patient with regulatory authority or private patient freedom

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-09 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study will be to compare the duration of post surgery hospitalisation between the patients who benefit with an alcohol weaning and the patient treated with usual methods. | two weeks
  time between the surgery and the exit of the hospital

SECONDARY OUTCOMES:
The secondary objective is to note: the presence of weaning syndrome, the diagnostic of Delirium tremens, the occurrence of post surgeries complications. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Albert TRAN, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Fédération des maladies de l'appareil digestif - Hôpital ARCHET, Nice, France